CLINICAL TRIAL: NCT02785653
Title: Effect of Sevoflurane on the Onset Characteristics and Intubating Conditions of Rocuronium Under Routine Clinical Practice
Brief Title: Effect of Sevoflurane on the Onset Characteristics and Intubating Conditions of Rocuronium
Acronym: SRI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maharashtra University of Health Sciences (Other)
Collaborators: Jaslok Hospital and Research Centre (Other)
Responsible Party: Principal Investigator, Nazmeen Sayed, Assistant Professor ,Department of Anaesthesia,Lokmanya Tilak Municipal Medical College and Hospital, Maharashtra University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR/ANAES/C/61
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Muscle Relaxation Caused by Sevoflurane
Keywords: sevoflurane; rocuronium; intubation
MeSH Terms: interventions — Sevoflurane; Rocuronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sevoflurane and rocuronium (Experimental): After induction of general anaesthesia, patients in the sevoflurane group were ventilated with fresh gas flow of 5 lites per minute consisting of 66.6% nitrous oxide and 33.3% oxygen with 2% inspired concentration of sevoflurane. After stabilization of end tidal carbondioxide to 30-35 mmHg ,intravenous rocuronium 0.6mg per Kg body weight was injected
  Interventions: Drug: Sevoflurane; Drug: Rocuronium
- rocuronium (Active Comparator): After induction of general anaesthesia, patients in the control group were ventilated with fresh gas flow of 5 lites per minute consisting of 66.6% nitrous oxide and 33.3% oxygen . After stabilization of end tidal carbondioxide to 30-35 mmHg ,intravenous rocuronium 0.6mg per Kg body weight was injected
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Sevoflurane — Patients were ventilated with 2 % inspired concentration of sevoflurane in a fresh gas flow of 5 litres containing 66.6% nitrous oxide and 33.3% percent of oxygen
  Other Names: Sevorane
  Arms: sevoflurane and rocuronium
Drug: Rocuronium — rocuronium 0.6mg per kg body weight was given intravenously after induction of anaesthesia
  Other Names: Esmeron

SUMMARY:
This study evaluates the potentiation of muscle relaxation caused by rocuronium by inhalational agent sevoflurane. Half the patients will be ventilated with oxygen ,nitrous oxide and sevoflurane during induction of anaesthesia and half will be ventilated only with oxygen and nitrous oxide.

DETAILED DESCRIPTION:
Rocuronium is a non depolarizing muscle relaxant. Inhalational general anaesthetic agents like Sevoflurane have some muscle relaxation effect by depressing the spinal motor neurons. Inhalational anaesthetics also alter the tonic input received from descending modulatory systems from the brain. Deep anaesthesia with inhalational agents may cause some degree of neuromuscular blockade.

ELIGIBILITY:
Inclusion Criteria:

* American society of anaesthesiologists physical status 1 and 2
* Age between 18-65
* Mallampatti classification 1 and 2

Exclusion Criteria:

* Patients refusal to participate
* American society of anaesthesiologists physical status 3 and 4
* Mallampatti classification 3 and 4
* Patients with neuromuscular disorder
* Patients on medications that affect neuromuscular block
* Pregnant and lactating patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
intubating condition | 10 minutes
  Copenhagen Consensus Conference Scale-scale to assess ease of intubation consisting of 5 parameters.laryngoscopy,vocal cord movement,vocal cord position,movement at intubation,coughing at intubation all are judged as poor ,good or excellent.If any parameter has a poor score, it is a clinically unacceptable intubating condition.

SECONDARY OUTCOMES:
lag time | 10 minutes
  time from start of rocuronium injection to first change in single twitch height on neuromuscular monitor
onset time for maximum relaxation | 10 minutes
  time from start of rocuronium injection to the disappearance of all four twitches on train of four stimulus on neuromuscular monitor

CONTACTS AND LOCATIONS:
Overall Officials: Nazmeen I Sayed, DNB(Anaes), Principal Investigator — Lokmanya Tilak Municipal Medical College and Hospital; Dipankar Dasgupta, MD(Anaes), Study Director — Jaslok Hospital and Research Centre
Locations (1):
- Jaslok Hospital and Research Centre, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No